CLINICAL TRIAL: NCT00915317
Title: Effect of Vitamin D Supplementation on Erythropoietin Dosage in Hemodialysis Patients Who Have Vitamin D Deficiency
Status: Withdrawn | Type: Observational
Why Stopped: Before we could start the study, we realized that many of the patients were already getting ergocalciferol. Therefore, the study was closed.
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 5125
Record Dates: First submitted 2008-10-15; First posted 2009-06-08 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Vitamin D Deficiency; Anemia
MeSH Terms: conditions — Vitamin D Deficiency; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
While vitamin D supplementation is safe and effective in repleting vitamin D levels in dialysis patients, the impact on anemia is unknown. The majority of hemodialysis patients require erythropoietin supplementation to maintain their serum hemoglobin between 11 and 12 gm/dL, a drug that is both costly and associated with significant side effects. If repletion of vitamin D significantly decreases erythropoietin requirements in hemodialysis patients, it would result in a substantial reduction in patient care costs. Our aim is to study the impact of ergocalciferol supplementation in hemodialysis patients with 25-hydroxyvitamin D deficiency. The investigators anticipate approximately 30% reduction in erythropoietin dose requirement in our hemodialysis population.

ELIGIBILITY:
Inclusion Criteria:

* All hemodialysis patients at the Kaiser Permanente Los Angeles Medical Center with vitamin D deficiency [defined by 25-hydroxyvitamin D level less than 30 ng/ml]

Exclusion Criteria:

* Non-renal causes of anemia (myelodysplastic syndrome, multiple myeloma, pure red cell aplasia, thallassemia, and sickle cell anemia)
* Active cancer
* AIDS
* refused erythropoeitin, intravenous iron or vitamin D analogs in the past
* no erythropoeitin requirement for greater than 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hemodialysis patients at the Kaiser Permanente Los Angeles Medical Center with vitamin D deficiency [defined by 25-hydroxyvitamin D level less than 30 ng/ml].
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
erythropoietin dosage | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Phillip S Yang, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Southern California, Los Angeles, California, United States

REFERENCES:
- [Background] Al-Aly Z, Qazi RA, Gonzalez EA, Zeringue A, Martin KJ. Changes in serum 25-hydroxyvitamin D and plasma intact PTH levels following treatment with ergocalciferol in patients with CKD. Am J Kidney Dis. 2007 Jul;50(1):59-68. doi: 10.1053/j.ajkd.2007.04.010. PMID 17591525
- [Background] Coen G, Mantella D, Manni M, Balducci A, Nofroni I, Sardella D, Ballanti P, Bonucci E. 25-hydroxyvitamin D levels and bone histomorphometry in hemodialysis renal osteodystrophy. Kidney Int. 2005 Oct;68(4):1840-8. doi: 10.1111/j.1523-1755.2005.00603.x. PMID 16164662
- [Background] Del Valle E, Negri AL, Aguirre C, Fradinger E, Zanchetta JR. Prevalence of 25(OH) vitamin D insufficiency and deficiency in chronic kidney disease stage 5 patients on hemodialysis. Hemodial Int. 2007 Jul;11(3):315-21. doi: 10.1111/j.1542-4758.2007.00186.x. PMID 17576296
- [Background] DeVille J, Thorp ML, Tobin L, Gray E, Johnson ES, Smith DH. Effect of ergocalciferol supplementation on serum parathyroid hormone and serum 25-hydroxyvitamin D in chronic kidney disease. Nephrology (Carlton). 2006 Dec;11(6):555-9. doi: 10.1111/j.1440-1797.2006.00698.x. PMID 17199797
- [Background] Ghazali A, Fardellone P, Pruna A, Atik A, Achard JM, Oprisiu R, Brazier M, Remond A, Moriniere P, Garabedian M, Eastwood J, Fournier A. Is low plasma 25-(OH)vitamin D a major risk factor for hyperparathyroidism and Looser's zones independent of calcitriol? Kidney Int. 1999 Jun;55(6):2169-77. doi: 10.1046/j.1523-1755.1999.00480.x. PMID 10354266
- [Background] Gonzalez EA, Sachdeva A, Oliver DA, Martin KJ. Vitamin D insufficiency and deficiency in chronic kidney disease. A single center observational study. Am J Nephrol. 2004 Sep-Oct;24(5):503-10. doi: 10.1159/000081023. Epub 2004 Sep 22. PMID 15452403
- [Background] LaClair RE, Hellman RN, Karp SL, Kraus M, Ofner S, Li Q, Graves KL, Moe SM. Prevalence of calcidiol deficiency in CKD: a cross-sectional study across latitudes in the United States. Am J Kidney Dis. 2005 Jun;45(6):1026-33. doi: 10.1053/j.ajkd.2005.02.029. PMID 15957131
- [Background] Martins D, Wolf M, Pan D, Zadshir A, Tareen N, Thadhani R, Felsenfeld A, Levine B, Mehrotra R, Norris K. Prevalence of cardiovascular risk factors and the serum levels of 25-hydroxyvitamin D in the United States: data from the Third National Health and Nutrition Examination Survey. Arch Intern Med. 2007 Jun 11;167(11):1159-65. doi: 10.1001/archinte.167.11.1159. PMID 17563024
- [Background] Saab G, Young DO, Gincherman Y, Giles K, Norwood K, Coyne DW. Prevalence of vitamin D deficiency and the safety and effectiveness of monthly ergocalciferol in hemodialysis patients. Nephron Clin Pract. 2007;105(3):c132-8. doi: 10.1159/000098645. Epub 2007 Jan 16. PMID 17228173
- [Background] Shah N, Bernardini J, Piraino B. Prevalence and correction of 25(OH) vitamin D deficiency in peritoneal dialysis patients. Perit Dial Int. 2005 Jul-Aug;25(4):362-6. PMID 16022093
- [Background] Taskapan H, Ersoy FF, Passadakis PS, Tam P, Memmos DE, Katopodis KP, Ozener C, Akcicek F, Camsari T, Ates K, Ataman R, Vlachojannis JG, Dombros NA, Utas C, Akpolat T, Bozfakioglu S, Wu G, Karayaylali I, Arinsoy T, Stathakis CP, Yavuz M, Tsakiris DJ, Dimitriades AD, Yilmaz ME, Gultekin M, Oreopoulos DG. Severe vitamin D deficiency in chronic renal failure patients on peritoneal dialysis. Clin Nephrol. 2006 Oct;66(4):247-55. doi: 10.5414/cnp66247. PMID 17063991
- [Background] Wolf M, Shah A, Gutierrez O, Ankers E, Monroy M, Tamez H, Steele D, Chang Y, Camargo CA Jr, Tonelli M, Thadhani R. Vitamin D levels and early mortality among incident hemodialysis patients. Kidney Int. 2007 Oct;72(8):1004-13. doi: 10.1038/sj.ki.5002451. Epub 2007 Aug 8. PMID 17687259
- [Background] Zadshir A, Tareen N, Pan D, Norris K, Martins D. The prevalence of hypovitaminosis D among US adults: data from the NHANES III. Ethn Dis. 2005 Autumn;15(4 Suppl 5):S5-97-101. PMID 16315387
- [Background] Zisman AL, Hristova M, Ho LT, Sprague SM. Impact of ergocalciferol treatment of vitamin D deficiency on serum parathyroid hormone concentrations in chronic kidney disease. Am J Nephrol. 2007;27(1):36-43. doi: 10.1159/000098561. Epub 2007 Jan 11. PMID 17215573